CLINICAL TRIAL: NCT03418337
Title: Comparison of the Efficiency of Two Different PPI Formula in Treatment of Atypical GERD Patients, a Randomized Study
Brief Title: Comparison of the Efficiency of Two Different PPI Formula in Atypical GERD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal Investigator (and Clinical Professor), Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-07-005A
Record Dates: First submitted 2018-01-18; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Compare the Response Rate of Atypical GERD After PPI Therapy
Keywords: cough, dexlansoprazole, GERD, globus, non-cardiac chest pain
MeSH Terms: conditions — Cough; Gastroesophageal Reflux; Globus Sensation | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Intervention Model Description: a prospective, randomized, open-level clinical study to evaluate 8 weeks PPI response rate for atypical GERD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexilansoprazole group (Dexilant 60 mg) (Experimental): After randomization, 60 subjects will receive oral dexlansoprazole (Dexilant 60 mg, Takeda Co. Ltd, Tokyo, Japan) once daily before breakfast for 8 weeks. Subjects will record their symptoms (cough, globus, NCCP, heart burn, and acid regurgitation) at daytime and nighttime everyday for 8 weeks. Symptoms suspecting drug adverse effect including nausea, diarrhea, constipation, headache, dizziness, fatigue, flatulence, etc will be recorded for 8 weeks.
  Interventions: Drug: dexilansoprazole (Dexilant 60 mg)
- lansoprazole group (Takepron OD 30 mg) (Active Comparator): After randomization, 60 subjects will receive oral lansoprazole (Takepron OD 30 mg, Takeda Co. Ltd, Tokyo, Japan) once daily before breakfast for 8 weeks. Subjects will record their symptoms (cough, globus, NCCP, heart burn, and acid regurgitation) at daytime and nighttime everyday for 8 weeks. Symptoms suspecting drug adverse effect including nausea, diarrhea, constipation, headache, dizziness, fatigue, flatulence, etc will be recorded for 8 weeks.
  Interventions: Drug: lansoprazole (Takepron OD 30 mg)

INTERVENTIONS:
Drug: dexilansoprazole (Dexilant 60 mg) — evaluate the response rate (symptom free) during the 8-week PPI therapy for atypical GERD between dexlansoprazole group and lansoprazole group
  Arms: dexilansoprazole group (Dexilant 60 mg)
Drug: lansoprazole (Takepron OD 30 mg) — lansoprazole group
  Arms: lansoprazole group (Takepron OD 30 mg)

SUMMARY:
Patients with atypical gastro-esophageal reﬂux disease (GERD), include cough, globus, and non-cardiac chest pain (NCCP) usually require more aggressive or double dose proton pump inhibitor (PPI) therapy than patients with typical GERD. Dexlansoprazole is a new, dual delayed release formulation of PPI that increases the mean intragastric pH during a 24-hour period. The prospective, open-label, randomized study aims to compare the efficacy of two different PPI formula in treating patients with atypical GERD symptoms.

Patients with atypical GERD symptoms and a total Reflux Symptom Index (RSI) score ≥13 (cough, globus, and NCCP) will be invited to participate. Personal characteristics including age, sex, body mass index, and the severity of erosive esophagitis will be recorded. After enrollment, 120 subjects will randomly assign (at a 1:1 ratio) to receive either oral lansoprazole, Takepron OD 30 mg, once daily before breakfast or oral dexilansoprazole, Dexilant 60 mg, once daily before breakfast for 8 weeks. Subjects will record their symptoms (cough, globus, NCCP, heart burn, and acid regurgitation) at daytime and nighttime everyday via diary for 8 weeks. The primary endpoint is to compare the cumulated incidence of each symptom free during 8-week therapy period between the two study groups. The secondary endpoint will be the withdrawal or drop-out rate due to poor symptoms response or drug adverse effects.

Data will be analyzed with SPSS Statistical Software for descriptive statistics (percentage, mean, standard error, and 95% confidence interval) and analytical statistics (chi-square test, ANOVA, and generalized estimation equation; GEE).

DETAILED DESCRIPTION:
We conduct a prospective randomized study since July 2017 after IRB approval. Patients between the ages of 20 and 80 years presenting to the gastroenterology outpatient clinic for atypical GERD symptoms (cough, globus, and NCCP) with or without typical symptoms (heartburn or acid regurgitation) of GERD will be invited to participate. After signing informed consents and screening, patients with atypical GERD symptoms for more than one month and with a total Reflux Symptom Index (RSI) score ≥13 were eligible for enrollment.Patients who currently took pro-kinetic agents, baclofen, antacid, sucralfate, histamin-2 receptor antagonists, PPI, antitussive, non-steroid anti-inflammatory drugs, anxiolytics, or anti-depressants or takes aforementioned medication during study period, who have severe cardiac, pulmonary, hepatic, or renal disease, who have uncured underlying malignancy, will be excluded as are subjects with laryngeal or pharyngeal disorders, a history of gastrointestinal (GI) surgery, symptoms of GI tract obstruction, or a contraindication for PPI use.

Personal characteristics including age, sex, habit of drinking and smoking, body mass index (BMI), waist circumference and underlying co-morbidity including diabetes, hypertension and dyslipidemia will be recorded. The findings of esophageal gastroduodenal scopy (EGD) will be recorded including the severity of erosive esophagitis (Los Angeles grade A-D or non-erosive reflux disease).The symptoms of atypical GERD including cough, globus sensation, and NCCP and the symptoms of typical GERD (heart burn and acid regurgitation) will be recorded everyday (daytime and night respectively) via diary before PPI therapy for 2 days and after PPI therapy for 8 weeks. The definitions of cough, globus sensation, NCCP, heart burn, and acid regurgitation will be according to a previous publication After enrollment, 120 subjects will randomly assign (at a 1:1 ratio) to receive either oral lansoprazole (Takepron OD 30 mg, Takeda Co. Ltd, Tokyo, Japan) once daily before breakfast or oral dexilansoprazole (Dexilant 60 mg, Takeda Co. Ltd, Tokyo, Japan) once daily before breakfast for 8 weeks. Subjects will record their symptoms (cough, globus, NCCP, heart burn, and acid regurgitation) at daytime and nighttime everyday for 8 weeks. Symptoms suspecting drug adverse effect including nausea, diarrhea, constipation, headache, dizziness, fatigue, flatulence, etc will be recorded for 8 weeks. Head elevation during sleeping, or on diet for body weight reduction, medication with pro-kinetic agents, baclofen, antacid, sucralfate, histamin-2 receptor antagonists, other PPI, antitussive, non-steroid anti-inflammatory drugs, anxiolytics, or anti-depressants will not be allowed during study period.

Endpoints We will evaluate the response rate (symptom free) everyday during the 8-week PPI therapy for cough, globus sensation, NCCP, acid regurgitation, and heartburn respectively. The primary endpoint is to compare the cumulated incidence and the time of each symptom free during 8-week therapy period between the two study groups. The secondary endpoint will be the withdrawal or drop-out rate due to poor symptoms response or drug adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. atypical GERD symptoms (cough, globus, or NCCP)
2. with or without typical GERD symptoms (heartburn or acid regurgitation)
3. A total Reflux Symptom Index (RSI) score ≥13

Exclusion Criteria:

1. Patients who currently took pro-kinetic agents, baclofen, antacid, sucralfate, histamin-2 receptor antagonists, PPI, antitussive, non-steroid anti-inflammatory drugs, anxiolytics, or anti-depressants during screening and during study period
2. Patients who have severe cardiac, pulmonary, hepatic, or renal diseases
3. Patients who have uncured underlying malignancy
4. Patients with laryngeal or pharyngeal disorders
5. Patients with a history of gastrointestinal (GI) surgery, symptoms of GI tract obstruction
6. Patients with a contraindication for PPI use

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The response rate of atypical GERD symptom | 8 weeks
  evaluate the response rate (symptom free) everyday during the 8-week PPI therapy for cough, globus sensation, NCCP, acid regurgitation, and heartburn respectively

SECONDARY OUTCOMES:
the withdrawal or drop-out rate between the two study groups | 8 weeks
  the withdrawal or drop-out rate due to poor symptoms response or drug adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided